CLINICAL TRIAL: NCT06668467
Title: The Effect of Mindfulness-Based Stress Reduction on Maternal Perceived Milk Supply: A Randomized Controlled Trial
Brief Title: The Effect of Mindfulness-Based Stress Reduction on Maternal Perceived Milk Supply
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19.04.2023/59
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breastfeeding
Keywords: Breastfeeding self-efficacy; Mindfulness; Insufficient milk; Social support; Stress
MeSH Terms: conditions — Breast Feeding | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Women assigned to the experimental group will receive mindfulness-based stress reduction training for 4 weeks.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Control (No Intervention): Women assigned to the control group will receive routine postpartum care services provided in the same hospital's outpatient clinics.

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — An 4-week Mindfulness-based stress reduction training programme
  Arms: Experimental

SUMMARY:
The aim of this study was to evaluate the effects of a mindfulness-based stress reduction (MBSR) programme on breastfeeding self-efficacy, stress, depression, anxiety and breastfeeding awareness in women with perceived breast milk insufficiency.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effects of a mindfulness-based stress reduction (MBSR) programme on breastfeeding self-efficacy, stress, depression, anxiety and breastfeeding awareness in women with perceived breast milk insufficiency.

The study is designed as a single-blind, randomised controlled trial. It will be conducted between November 2024 and January 2025 at the Zeynep Kamil Women and Children's Diseases Education and Research Hospital.

Power analysis using G*Power showed that at least 35 samples would be sufficient for 2 groups with an effect size of 0.5, 95% power and 5% margin of error. Participants to be included in the groups were selected from the sample using a random sampling method with an equal distribution ratio (distribution ratio = 1:1).

Eligible women were randomised to the intervention group (n=35) and the control group (n=35). Women allocated to the intervention group received the MBSR programme. MBSR was scheduled for 4 weekly sessions of 30 minutes each. The control group received routine hospital care but no other intervention during this period.

The pre-test data for the study were collected by the researcher using face-to-face interviews, a personal information form with demographic questions and the measurement tools used in the study. After one week and at the end of 4 weeks, the same measurement tools were used to collect post-test data.

Participants were given information about the MBSR programme and told how, for how long, and where they would practise. The online MBSR programme was completed by the participants in a specific way for each session (with mind, body and breathing exercises). The MBSR programme was delivered in this way for 4 weeks (eight sessions in total, two sessions per week). In addition, participants were given homework (audio recordings) to repeat the mindfulness meditation practices throughout the week (until the next session). At the end of the fourth week, the measures were administered again to participants who had attended all eight sessions and completed their homework, and post-test data were collected.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* 37 weeks or more of gestation
* Primipar
* Having given birth vaginally
* University Health Application and Research Center, Gynaecology and Obstetrics Clinic
* Having a single and healthy baby (no multiple pregnancy)
* Having completed at least primary school
* Being able to communicate in Turkish by phone using the WhatsApp application
* The baby is with the mother

Exclusion Criteria:

* Having a high-risk pregnancy
* Having a medical condition or taking medication that prevents breastfeeding
* Having a communication problems (vision, hearing, speech, language problems)
* Having a psychiatric illness
* There is an obstacle that prevents the baby from being with the mother or being in the neonatal intensive care unit
* Having a condition/disease that prevents you from doing mindfulness practices (breathing exercises, body scanning)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Famale
Enrollment: 100 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Mindful Breastfeeding Scale (MIND-BFS) | Day 1, Day 7, Day 30 after delivery
  The Mindful Breastfeeding Scale (MIND-BFS) is a 9-item measurement tool that evaluates awareness-based breastfeeding practices in the postpartum period. The scale is one-dimensional and was developed as a 5-point Likert type. Responses to the scale items vary from (1) Always to (5) Never. The total score to be obtained from the scale is scored between 9-45, and as the total score obtained from the scale increases, the awareness rate of breastfeeding also increases.
Breastfeeding Self-Efficacy Scale | Day 1, Day 7, Day 30 after delivery
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed. The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short form was performed by Aluş Tokat and Okumus in 2009. This scale assesses how competent mothers feel about breastfeeding. The scale consists of 14 items and includes a 5-point Likert-type evaluation consisting of Not sure at all: 1, Not very sure: 2, Sometimes I am sure: 3, I am sure: 4, Very sure: 5 options. The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy.
Depression, Anxiety and Stress Scale (DASS-21) | Day 1, Day 7, Day 30 after delivery
  The scale consists of 21 items and three sub-dimensions. Each of the seven items that make up each sub-dimension of the scale measures depression, anxiety and stress. The DASS-21 scale is a four-point Likert-type scale and the items are evaluated between 0 and 3 (0 = not at all suitable for me, 1 = somewhat appropriate for me, 2 = usually suitable for me, 3 = completely suitable for me). There is no reverse item in the scale. The total scores of the scale range from 0 to 21 for each sub-dimension. In the validity and reliability study, the Cronbach-alpha coefficient was determined as 0.87 for the depression sub-dimension, 0.85 for the anxiety sub-dimension, and 0.81 for the stress sub-dimension. The Cronbach-alpha coefficient for the Turkish version of the Depression, Anxiety and Stress scale was determined as 0.88 for the depression sub-dimension, 0.80 for the anxiety sub-dimension and 0.87 for the stress sub-dimension
Multidimensional Scale of Perceived Social Support (MSPSS) | Day 1, Day 7, Day 30 after delivery
  MSPSS is a 12-item scale that measures the adequacy of social support. It consists of 3 subgroups that include items about family, friends and social support from a special person. It consists of 4 items for each group and each item is graded on a 7-item likert scale. A high total score indicates a high level of perceived social support.
Insufficient Milk Perception Scale | Day 1, Day 7, Day 30 after delivery
  The Insufficient Milk Perception Scale is a scale developed by McCarterSpaulding (2001) to measure mothers' beliefs about whether they produce sufficient milk. It consists of 6 questions. A minimum score of 0 and a maximum score of 50 can be obtained from this scale. A high score indicates that the mother's perception of adequate milk is high

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kaya, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)